CLINICAL TRIAL: NCT06557278
Title: Phase II Open-Label Study to Assess the Safety and Efficacy of AlloStim® + Anti-PDL1 as Fourth Line Therapy in 4L MSS Metastatic Colorectal Cancer
Brief Title: Combined AlloStim+Anti-PD-L1 in 4L MSS Metastatic Colorectal Cancer
Acronym: COMUNITY
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Redesign of protocol for primary end-point of overall survival
Sponsor: Mirror Biologics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MBI-006-COMUNITY
Record Dates: First submitted 2024-08-08; First posted 2024-08-16 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Colorectal Cancer
Keywords: colorectal cancer; checkpoint inhibitor; AlloStim; immunotherapy; avelumab
MeSH Terms: conditions — Colorectal Neoplasms | interventions — avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Biological: AlloStim — experimental immunotherapy to prime for checkpoint inhibitor
Drug: Bavencio — anti-PDL1 checkpoint inhibitor
  Other Names: Avelumab

SUMMARY:
Experimental immunotherapy in chemotherapy-refractory and immunotherapy-refractory metastatic colorectal cancer patients that have progressed, or are intolerant to, Longsurf (TAS-102) +/- Avastin (bevacizumab) or Stivarga (regorafenib) or Fruzaqla (fruquintinib) combining experimental AlloStim with an anti-programmed death ligand 1 (PD-L1) checkpoint inhibitor drug.

DETAILED DESCRIPTION:
The protocol provides fourth-line experimental treatment for subjects with microsatellite stable (MSS)/ proficient mismatch repair (pMMR) metastatic colorectal cancer. These patients do not respond to checkpoint inhibitors. This study will investigate whether AlloStim® administered weekly in two-21 day cycles with each cycle consisting of 3 weekly intradermal (ID) doses followed the last week with an intravenous (IV) dose (3 cycles =Days 0 through 49) can prime patients to become responsive to checkpoint inhibition immunotherapy. A restaging computed tomography (CT) scan is conducted on day 56 after the priming and will be compared to the baseline CT scan by Response Evaluation Criteria in Solid Tumors (RECIST 1.1). Scans at day 56 are expected to be read as radiological progression upon restaging after AlloStim® priming, possibly due to immunological swelling, known as "pseudoprogression", consistent with the presumed inflammatory mechanism of action of AlloStim®. This mechanism may convert "cold" tumors to "hot" tumors. The immune cell infiltrates of tumors after AlloStim® include T-helper cell type 1 (Th1) memory cells which produce interferon-gamma. Interferon-gamma is known to increase expression of anti-programmed death ligand 1 (PD-L1) checkpoint molecules in the tumor microenvironment. Higher PD-L1 expression may convert checkpoint inhibitor unresponsive tumors to become checkpoint inhibitor responsive. After two 21-day cycles of AlloStim® priming, a combination of AlloStim® IV boosters and anti-PD-L1 checkpoint therapy (with avelumab 800 mg q/2 weeks) is scheduled between days 63 to day 98, A restaging CT scan at day 112 is then compared to day 56 and baseline to determine if the tumor target lesions' size has changed. An expansion phase providing another cycle of combined AlloStim® and avelumab is provided for stable patients from days 119-154. A final restaging CT scan is conducted on Day 168 for all subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male and female subjects aged 18-80 years at screening visit
2. Pathologically confirmed diagnosis of MSS/pMMR colorectal adenocarcinoma
3. Presenting with metastatic disease:

   * Primary tumor can be intact or previously resected
4. Previous treatment failure of at least two lines of active systemic chemotherapy:

   * Previous chemotherapy must have included a fluoropyrimidine, oxaliplatin (e.g. FOLFOX, CAPOX), and irinotecan-containing (e.g. FOLFIRI) regimens (single regimen of FOLFIRINOX satisfies)
   * Administered in adjuvant setting or for treatment of metastatic disease
   * If KRAS wild type, must have at least one prior anti-EGFR therapy if left sided primary tumor
5. Treatment failure or refusal/not qualified for at least one third-line treatment

   * TAS-102 +/- bevacizumab or regorafenib or fruquinib
   * Treatment failure can be due to disease progression or toxicity
   * Time from last treatment failure to Informed Consent must be no more than 30 days
6. ECOG performance score: 0-1
7. Adequate hematological function:

   * Absolute granulocyte count ≥ 1,200/mm3
   * Platelet count ≥ 100,000/mm3
   * Hemoglobin ≥ 9.0 g/dL (may be corrected by transfusion)
8. Adequate Organ Function:

   * Creatinine ≤ 1.5 mg/dL
   * Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
9. Alkaline phosphatase ≤ 2.5 times ULN *
10. Aspartate aminotransferase (AST) or (SGOT) ≤ 2.5 times ULN *
11. Alanine aminotransferase (ALT) or (SGPT) ≤ 2.5 times ULN*
12. EKG without clinically relevant abnormalities
13. Female subjects: Not pregnant or lactating
14. Patients with childbearing potential must have a negative ß-HCG test and agree to use a highly effective contraceptive method during the course of the study
15. Study specific Informed Consent in the native language of the subject

    * ≤ 5 times ULN if liver involvement

Exclusion Criteria:

1. High frequency microsatellite instability (MSI-H) or deficient mismatched repair dMMR
2. Bowel obstruction or high risk for obstruction if tumors become inflamed
3. Moderate or severe ascites requiring medical intervention
4. Clinical evidence of brain metastasis or leptomeningeal involvement
5. Widespread peritoneal carcinomatous (e.g. CT scan shows innumerable lesions visible and/or abnormal thickening of greater omentum) that increases risk of a major morbidity (e.g. bowel obstruction) in the opinion of the Investigator
6. COPD
7. Pulmonary lymphangitis or symptomatic pleural effusion (grade ≥ 2) that results in pulmonary dysfunction requiring active treatment; or, oxygen saturation <92% on room air
8. Any of the following mood disorders: active major depressive episode, recent history of suicidal attempt or ideation
9. Prior allogeneic bone marrow/stem cell or solid organ transplant
10. Chronic use (> 2 weeks) of greater than physiologic doses of a corticosteroid agent (dose equivalent to > 5 mg/day of prednisone) planned or anticipated during the study before the end of the Safety Evaluation Period (28 days after the last dose of IP)

    * Topical corticosteroids are permitted
11. Prior diagnosis of an active autoimmune disease (e.g., rheumatoid arthritis, multiple sclerosis, autoimmune thyroid disease, uveitis)

    * Well controlled Type I diabetes allowed (HbA1c < 8.5%)
12. Prior experimental immunotherapy
13. History of blood transfusion reactions
14. Progressive viral or bacterial infection

    o All infections must be resolved and the subject must remain afebrile for seven days without antibiotics prior to being placed on study
15. Cardiac disease of symptomatic nature
16. History of HIV positivity or AIDS
17. History of severe hypersensitivity to monoclonal antibody drugs
18. Psychiatric or addictive disorders or other condition that, in the opinion of the Investigator, would preclude study participation.
19. Subjects that lack ability to provide consent for themselves
20. Any prior cancer diagnosis (other than cured basal cell carcinoma, head and neck carcinoma in-situ, superficial Ta, Tis, T1 bladder cancer, or papillary carcinoma of thyroid) or concurrent cancer histologically different than colorectal adenocarcinoma

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-11 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Objective Tumor Response | day 168
  CT scan RESIST 1.1
Overall Survival | 2 years
  survival from signing consent until death by any cause

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Mt. Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Hirschfield Oncology Center, Brooklyn, New York
  - New York Cancer and Blood Specialists, Shirley, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Case Report — https://rdcu.be/dHXGN